CLINICAL TRIAL: NCT00137592
Title: Promoting Colorectal Cancer Screening in Rural Colorado
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-4547; PRC SIP 20-04
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer
Keywords: screening; community health education
MeSH Terms: conditions — Colorectal Neoplasms; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Experimental): Behavioral: small media, group education (multicomponent)
  Interventions: Behavioral: small media, group education (multicomponent)

INTERVENTIONS:
Behavioral: small media, group education (multicomponent)

SUMMARY:
This community based participatory research study involves multicomponent educational interventions. Telephone interviews and focus groups of persons who are residents of the High Plains region of Colorado will be conducted. A card study will also be carried out to collect limited data about colorectal cancer screening in primary care practices. The multicomponent intervention approaches (e.g., small media and group education) consist of educational materials about routine colorectal cancer screening.

DETAILED DESCRIPTION:
Specific Aims:

* Using community-based participatory research (CBPR), incorporate an existing Community Advisory Council into a project-specific Joint Planning Committee to provide community voices and be experts for a project to design strategies to improve CRC screening of all adults over the age of 50 in the High Plains community.
* Work with the Joint Planning Committee to develop an acceptable and respectful message and dissemination plan to change the community perception concerning colorectal cancer screening.
* Conduct a random digit dialing survey of rural eastern Colorado to determine rates of individuals up to date on CRC screening and to determine current knowledge level of individuals over 50 concerning the need for CRC screening.
* Deliver the screening message(s) through the methods suggested by the Joint Planning Committee in two High Plains communities and solicit community members' reactions to the message(s) and dissemination approaches.

Setting

The Intervention Communities:

The nine rural counties within northeast Colorado that make up the High Plains communities encompass 15,000-square-miles. The economy is largely agricultural, with a population of approximately 90,000. Based on the 2000 census 22% (range 20-29%) of the population is over 50, which is higher than the state as a whole (20%) or the Denver Metropolitan Statistical Area - MSA (18%). There is not a single MSA in the High Plains region and most of the region is a frontier area and therefore considered an underserved community.

The Control Communities:

We will also utilize the 8 county region in southeastern Colorado as our control communities for the intervention evaluation.

Primary Care Offices:

This study will be conducted within the community detailed above. The intervention will be at the population level. Evaluation of the intervention will include surveys of providers and patients within the primary care offices in the High Plains Region (these offices are part of the High Plains Research Network [HPRN]) and piloting the intervention will occur in the primary care practices that are part of the Colorado Research Network (CaReNet). Both CaReNet and HPRN are practice based research networks (PBRNs) affiliated with the Department of Family Medicine at the University of Colorado.

Project Aims (Overview):

We will combine three different proven research approaches to develop and study a community-based intervention to improve CRC screening rates.

- Component 1: Intervention Planning:

* Using a community-based participatory research model, the Joint Planning Committee (JPC) composed of members of an established Community Advisory Council for a practice-based research network and other community members, we will explore and define the messages and the delivery approaches the community members feel are most likely to result in actual behavioral change.

  * Component 2: Assessment of Intervention Effectiveness:
* Using a random digit dialing telephone survey, pre and post provider/patient card study and a provider survey, we will assess the impact of the intervention.

  * Component 3: Evaluation of Intervention Process and Implementation:
* Using the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework12, we will guide our evaluation of both the community-based participatory research process and the effects of the intervention developed.

ELIGIBILITY:
Exclusion Criteria:

* Colorectal cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
colorectal cancer screening | 30 days

SECONDARY OUTCOMES:
colorectal cancer screening knowledge | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: John M. Westfall, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States